CLINICAL TRIAL: NCT02592499
Title: Swedish Evaluation of Left Ventricular Assist Device
Brief Title: Swedish Evaluation of Left Ventricular Assist Device as Permanent Treatment in End-stage Heart Failure
Acronym: SweVAD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Vastra Gotaland Region (Other Government)
Collaborators: Karolinska University Hospital (Other); University Hospital, Linkoeping (Other); Skane University Hospital (Other); Uppsala University Hospital (Other); University Hospital, Umeå (Other); Region Örebro County (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: ver 6.0; 635-14 (Other: Sweden: Regional Ethical Review Board)
Record Dates: First submitted 2015-10-23; First posted 2015-10-30 (Estimated); Last update posted 2023-04-26 (Actual); Status verified 2023-04

CONDITIONS: End-stage Heart Failure
Keywords: HM III; survival; LVAD

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- HM III (Experimental): Patients randomized to mechanical circulatory support will be treated with the HeartMate III (HM III) left ventricular assist device system.
  Interventions: Device: HM III
- OMM, Optimal Medical Management (Active Comparator): Patients randomized to OMM will be treated according to international guidelines.
  ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure 2012: The Task Force for the Diagnosis and Treatment of Acute and Chronic Heart Failure 2012 of the European Society of Cardiology. Eur Heart J. 2012 Jul;33(14):1787-84
  Interventions: Other: OMM, optimal medical management

INTERVENTIONS:
Device: HM III
  Other Names: left ventrical assist device, LVAD
  Arms: HM III
Other: OMM, optimal medical management — Patients randomized to OMM will be treated according to international guidelines. All patients should receive a beta blocker, an ACE-inhibitor or an Angiotension II receptor blocker, and a mineralocorticoid receptor antagonist if tolerated and at optimally titrated doses according to guidelines. Loop diuretics should also be used as needed to control fluid retention. Other drugs that may relieve symptoms and improve prognosis can be used (incl ivabradin, digoxin, hydralazine,isosorbiddinitrate, anticoagulant agents). Patients that have an indication for implantable cardioverter defibrillator (ICD) and/or cardiac resynchronization therapy (CRT) should receive such therapy. Surgical interventions that may be indicated for specific underlying or contributing causes of heart failure.
  Arms: OMM, Optimal Medical Management

SUMMARY:
The study is a prospective, randomized, non-blinded, national, multi-center study. The study will consist of the assignment of eligible patients to treatment with either a HeartMate III (HM III) left ventricular assist device system or to pharmacological treatment (optimal medical management, OMM) according to current guidelines. Eighty (80) patients will be enrolled in this study and randomized in a 1:1 fashion between the HM III and OMM, based on a modified power calculation.

DETAILED DESCRIPTION:
The primary objective is to compare survival between left Ventricular Assist Device (LVAD) destination therapy and optimal medical management in a Swedish end stage heart failure population ineligible for cardiac transplantation.

The secondary objective is to compare treatment groups with respect to organ function, functional capacity, quality of life and adverse events.

All patients enrolled in the study will be followed through 2 years. Patients who continue to be on going with the HM III or on OMM past 2 years will continue be followed for their outcomes and adverse events for up to 5 years. Patient recruitment was expected to occur over 24 months, but due to difficulties in recruiting patients will be longer (approximately 48 months)

The study will be conducted in Sweden at all 7 University Hospitals and implantations will be performed in 5 sites.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent
2. Adult (≥ 18 years)
3. Chronic heart failure ≥ 45 days or stable not supported by mechanical circulatory support since >7days on single inotrope.
4. Left ventricular ejection fraction ≤ 30%.
5. NYHA IIIB-IV, INTERMACS profile 2-6
6. At least 2 of 4 adverse prognostic criteria:

   * SHFM estimated 1-year survival ≤75%
   * NTproBNP ≥ 2000 ng/l
   * VO2 max < 14 ml/kg/min or <50% of predicted VO2max with attainment of anaerobic threshold (AT), or unable to perform.
   * Need for continuous or intermittent inotropic support or >2 hospitalizations during last 6 months.
7. Receiving medical management with optimal doses of betablockers, ACE-inhibitors or ARBs, and MRAs for at least 30 days if tolerated.
8. Receiving CRT if indicated for at least 45 days.
9. Receiving ICD if indicated and appropriate.
10. Ineligible for cardiac transplantation (e.g. high age and/or co-morbidities)
11. Considered suitable for the study by a multidisciplinary board

Exclusion Criteria:

1. Eligible for heart transplantation or is likely to become eligible after VAD treatment (bridge-to-candidacy)
2. Indication for revascularisation, valvular surgery or other cardiac intervention expected to improve cardiac function and prognosis (CABG, PCI TAVI, mitraclip etc.)
3. INTERMACS profile 1 "crash and burn"
4. On-going mechanical circulatory support.
5. Heart failure due to restrictive cardiomyopathy pericardial disease, active myocarditis or uncorrected thyroid disease.
6. Mechanical aortic valve that will not be converted to a bioprosthesis or patch
7. Moderate to severe aortic insufficiency without plans for correction
8. Technical obstacles, which pose an inordinately high surgical risk
9. Active, uncontrolled infection

11. Stroke within 90 days or carotid artery stenosis > 80 % 12. Significant vascular disease. 13. Severe COPD or severe restrictive lung disease. 14. Intrinsic hepatic disease as defined by liver enzyme values (AST or ALT or total bilirubin) > 5 times the upper limit of normal, or INR > 2.0, which is not due to anti-coagulant therapy.

15. Intolerance to anticoagulant or antiplatelet therapies or any other operative therapy the patient will require based upon the patient's health status.

16. Platelet count < 50,000. 17. Measured GFR <20 ml/min/1.73m2 unresponsive to inotrope treatment or chronic dialysis.

18. High risk for right ventricular failure according to echocardiography and/or invasive hemodynamic measurements as judged by the investigator (>2 parameter constitute an exclusion criteria) using a combination of the:

a. Severe TI b. TAPSE < 0.72 cm c. RVEDD/LVEDD > 0.72 d. CVP > 16 mm Hg e. MPAP - RAP < 10 mmHg SPAP-DPAP/CVPm >1 ok, <0.5 very bad, in between borderline f. CVP/PCWP > 0.63 g. RVSWI < 300 mm Hg x ml/m2 h. Bilirubin > 34 micromol/L 19. Body Mass Index (BMI) > 42 kg/m2. 20. Psychiatric disease, cognitive dysfunction, alcohol or drug abuse, or psychosocial issues that are likely to impair study compliance 21. Female of childbearing age with a positive pregnancy test or not willing to use adequate contraceptive precautions during the study.

22. Condition, other than heart failure, that could limit survival to less than 2 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2016-06 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Survival at two years of follow-up | 2 years,
  survival

SECONDARY OUTCOMES:
Number of participants free from disabling stroke during the 2-year follow-up period | 2 years
  Survival free from disabling stroke (Modified Rankin Scale (MRS) >3)
A composite endpoint of "survival free from disabling stroke", survival and non-planned hospitalizations | 2 years
  Survival free from a composite endpoint of disabling stroke, survival and non-planned hospitalizations
Survival at year of follow-up | 1 year
  Survival at year
Functional capacity (NYHA) during the 2-year follow-up period | 2 years
  functional capacity determined by NYHA classification
Functional capacity (6 min walk-test) during the 2-year follow-up period | 2 years
  functional capacity determined by 6 min walk-test
Functional capacity (peak VO2) | 2 years
  functional capacity determined by peak VO2
Health-related quality of Life during the 2-year follow-up period | 2 years
  Health-related quality of Life asses with EQ-5D-5L, SF-36 and KCCQ
Number of participants with heart-failure related events | 2 years
Cost-effectiveness during the 2-year follow-up period | 2 years
  Cost effectiveness calculated with QUALY (Quality-adjusted Life-year) and LY (Life year)
Renal function during the 2-year follow-up period | 2 years
  Glomerular filtration rate evaluated by 51 chrome-EDTA or Iohexol clearance
Hospital admissions during the 2-year follow-up period | 2 years
  Number of hospital admissions
Number of participants with serious adverse events (SAEs) | 2 years
Functional capacity (peak VO2) | 1 year
  functional capacity determined by peak VO2
Three-years survival | 3 years
  survival
Four-years survival | 4 years
  survival
Five-years survival | 5 years
  survival

CONTACTS AND LOCATIONS:
Overall Officials: Kristjan Karason, MD, Principal Investigator — Vastra Gotaland Region
Locations (7):
- Sweden (7):
  - Sahlgrenska Univesitetssjukhustet, Transplantationscentrum, Gothenburg
  - Linköping Univ Hospital, Linköping
  - Skåne University Hospital, Lund
  - Örebro Univ Hospital, Örebro
  - Karolinska Univ Hospital, Stockholm
  - Univ Hospital of Umeå, Umeå
  - Uppsala Univ Hospital, Uppsala

IPD SHARING:
Plan to Share IPD: Yes
We have not yet made an exact plan but see no reason for not sharing the data regarding IPD underlying the results of the study, as well as the protocol, SAP and ICF after publication, but will also depend on requirement by the journal upon publication.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: After publication
Access Criteria: Not decided yet